CLINICAL TRIAL: NCT03712943
Title: Phase I Study of Regorafenib and Nivolumab in Mismatch Repair (MMR) Proficient Advanced Refractory Colorectal Cancer
Brief Title: Regorafenib and Nivolumab in Mismatch Repair (MMR) Refractory Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19581
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer; Colon Cancer
Keywords: colon cancer; colorectal; MMR; Mismatch Repair
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Regorafenib and Nivolumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Regorafenib and Nivolumab Combination - Escalation (Experimental): Dose Escalation: To find the dose of regorafenib that can be safely given with nivolumab in patients with advanced, refractory colorectal cancers.
  Interventions: Drug: Regorafenib; Drug: Nivolumab
- Regorafenib and Nivolumab Combination - Expansion (Experimental): Dose Expansion: To find the effect on tumor of the combination of regorafenib and nivolumab.
  Interventions: Drug: Regorafenib; Drug: Nivolumab

INTERVENTIONS:
Drug: Regorafenib — Regorafenib orally 80 mg daily for 21 days (3 weeks on, 1 week off).
  Other Names: Stivarga
Drug: Nivolumab — Nivolumab 240 mg administered intravenously every 2 weeks.
  Other Names: OPDIVO

SUMMARY:
The main purpose of this study is to test the safety, tolerable side effects, and determine the highest tolerable dose of the combination of Regorafenib and Nivolumab. Researchers want to find out if this combination of Regorafenib and Nivolumab can help people with metastatic colorectal cancer with mismatch repair (MMR) proficiency.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal adenocarcinoma
* Proficient DNA mismatch repair (MMR) or stable microsatellite disease.
* Participants with the presence of at least one lesion with measurable disease as defined by 10mm in longest diameter for a soft tissue lesions or 15mm in short axis for a lymph node by RECIST 1.1 for response assessment.
* Participants must have received and progressed through or become intolerant to fluoropyrimidine, irinotecan, oxaliplatin, and bevacizumab, and if K-ras wild type, cetuximab or panitumumab containing therapies. Exceptions may apply.
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1
* Estimated life expectancy over 3 months.
* Adequate bone marrow, liver and renal function.
* Participants must not have had chemotherapy, major surgery, monoclonal antibody therapy or experimental therapy within the 21 days prior to the start of regorafenib and nivolumab administration
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) performed within 24 hours prior to the start of study drug and then every 4 weeks. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Participants (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the Informed Consent Form (ICF) until at least 5 months for females and 7 months for males after the last dose of study drug
* Participants must be able to understand and be willing to sign the written informed consent form and be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.

Exclusion Criteria:

* Participants with active Central Nervous System (CNS) metastases If CNS metastases are treated and participants are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment.
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v5.0] on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease.
* Women who are pregnant or breast-feeding
* Prior therapy with regorafenib, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks
* Participants with phaeochromocytoma
* Ongoing infection > Grade 2
* Presence of a non-healing wound, or bone fracture.
* Renal failure requiring hemo-or peritoneal dialysis.
* Seizure disorder requiring medication.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Persistent proteinuria ≥ Grade 3
* History of organ allograft
* Participants requiring warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon)
* Participants with a condition requiring a strong CYP3A4 inhibitors or strong CYP3A4 inducers.
* Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy or procedure, excluding alopecia.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Participants with an arterial thrombotic or thromboembolic event within 6 months of informed consent.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection.
* Child-Pugh B cirrhosis (or worse) or a history of hepatic encephalopathy
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
* Participants requiring concurrent anti-cancer therapy other than study treatment.
* Participants requiring hormonal therapy during the study or within 2 weeks of first study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 12 months
  To determine the maximum tolerated dose of Regorafenib in combination with Nivolumab in advanced, refractory colorectal cancers.

SECONDARY OUTCOMES:
Response Rate | Every 2nd cycle (Cycles are 28 days) up to 12 months
  To access response rate using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Overall Survival (OS) | Up to 24 months after conclusion of treatment
  Occurrence of Overall Survival
Frequency and Severity of Adverse Events | Up to 12 months
  To evaluate the frequency and severity of adverse events and tolerability of the combination regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Dae W Kim, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Kim RD, Kovari BP, Martinez M, Xie H, Sahin IH, Mehta R, Strosberg J, Imanirad I, Ghayouri M, Kim YC, Kim DW. A phase I/Ib study of regorafenib and nivolumab in mismatch repair proficient advanced refractory colorectal cancer. Eur J Cancer. 2022 Jul;169:93-102. doi: 10.1016/j.ejca.2022.03.026. Epub 2022 May 5. PMID 35526308